CLINICAL TRIAL: NCT04956185
Title: Prospective Data Collection of Patients Admitted to the Stroke Unit At University Hospital Ghent
Brief Title: Data Collection of Patients Admitted to the Stroke Unit
Acronym: PRODA-STROKE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-09645
Record Dates: First submitted 2021-04-29; First posted 2021-07-09 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Stroke, Acute; Stroke, Ischemic; Stroke Hemorrhagic; Stroke Sequelae
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this prospective observational study is to create a database in which data will be collected from every patient admitted to the Stroke unit and who has explicitly given his or her informed consent for this data collection. The data that will be collected are part of the standard clinical data. No additional investigations, blood tests or any other tests will be performed. The purpose of this database is to conduct retrospective observational research in the future and will allow the hospital to keep track of some important quality indicators in stroke care.

DETAILED DESCRIPTION:
Every patient that is admitted to the Stroke unit will be asked if his or her data and relevant personal information can be registered in a database with the purpose of conducting research in the future. If he or she agrees, one of the researchers will go through the Informed Consent Form together with the patient. If the patient has questions, the researcher will answer them. If the patient then agrees to the data collection, he or she will sign the Informed Consent Form.

The data that will be collected are part of the standard clinical data. No additional investigations, blood tests or any other tests will be performed. We will collect the following data:

* Demographical information: gender, year of birth
* Relevant medical history: vascular risk profile, neurological history, psychiatric history, pre-stroke modified Rankin Score (mRS), home medication
* Neurological evaluation upon admission to Emergency Department: vital parameters, clinical neurological evaluation, results imaging
* Data concerning acute stroke therapy: intravenous thrombolysis, intra-arterial thrombectomy, medication started at the Emergency Department, neurosurgical procedures if performed, (neurological) evaluation after treatment
* Course of hospitalisation: complications (neurological deterioration, epilepsy, infections, falls, speech or swallow disturbances, thrombo-embolic complications, pain, cardiac complications), start of medication, treatment (such as physiotherapy, occupational therapy), date of discharge, mRS and NIHSS score at discharge, care after discharge
* Results stroke-investigations: imaging of brain and neck vessels, telemetry, Holter monitoring, transthoracic and/or transesophageal ultrasound, blood workup, electro-encephalographic investigations, genetic workup, etiology of stroke
* Therapy at discharge: medication, revalidation
* mRS score during follow-up at policlinic neurology

The purpose of this database is to conduct retrospective observational research in the future and will allow the hospital to keep track of some important quality indicators in stroke care.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Stroke unit with a cerebrovascular disease
* Patients admitted to the regular neurological ward or any other department in the University Hospital Ghent with a cerebrovascular disease who are actively followed by the department of Neurology during hospitalisation
* Patients who have given their explicit informed consent for data collection

Exclusion Criteria:

* Patients who have not given informed consent for data collection
* Patients who are not able to give informed consent and whose legal representative has not given informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to the Stroke unit (or to any other hospital ward) with a cerebrovascular disease and who have given their informed consent for data collection (or whose legal representative has given informed consent for data collection).
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2031-02-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Characteristics of study population | date of inclusion until end of follow-up (12 months)
  Information about patients included in the stroke database: age, gender, medical/family history
Onset-to-door | date of inclusiondate of inclusion until end of follow-up (12 months)
  Time between stroke onset and arrival at Emergency Department
Patients treated with acute stroke therapy | date of inclusion until end of follow-up (12 months)
  Patients treated with acute stroke therapy (i.e. thrombolysis and/or thrombectomy), start time of acute therapy
Outcome after acute therapy | date of inclusion until end of follow-up (12 months)
  Outcome after acute therapy, assessed by NIHSS and mRS score, possible complications and imaging
Incidence of complications at stroke unit | date of inclusion until end of follow-up (12 months)
  Incidence of neurological complications, epilepsy, infections, falls, thrombo-embolic complications, cardiac complications, pain
Etiology of stroke | date of inclusion until end of follow-up (12 months)
  Etiology of stroke, with a distinction between ischaemic stroke, hemorrhagic stroke, subarachnoid stroke or other
Mortality and disability after admission to Stroke unit | date of discharge until end of follow-up (12 months)
  Mortality and (severity of) disability after admission to stroke unit

SECONDARY OUTCOMES:
Quality of stroke care | date of inclusion until end of follow-up (12 months)
  Quality of care at Stroke unit of the University Hospital Ghent

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology - Ghent University Hospital, Ghent, Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No